CLINICAL TRIAL: NCT01248962
Title: Standard Infusion Carboplatin Versus Prophylactic Extended Infusion Carboplatin in theTreatment of Patients With Recurrent, Ovary, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Standard Infusion Carboplatin Versus Prophylactic Extended Infusion Carboplatin in Patients With Patients With Recurrent, Ovary, Fallopian Tube, and Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-184
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: BEVACIZUMAB (AVASTIN); CARBOPLATIN; DEXAMETHASONE; GEMCITABINE; LIPODOX(LIPOSOMAL DOXORUBICIN); MONTELUKAST (SINGULAR); TAXOL (PACLITAXEL; Fallopian Tubes; 10-184
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard 30-minute infusion (Experimental): This is a non-blinded randomized study comparing standard 30-minute infusion carboplatin to extended 3-hour infusion carboplatin in women with recurrent, ovary, fallopian tube, and primary peritoneal cancer who will be treated with a carboplatin containing chemotherapy regimen.
  Interventions: Drug: carboplatin
- extended 3-hour infusion (Experimental): This is a non-blinded randomized study comparing standard 30-minute infusion carboplatin to extended 3-hour infusion carboplatin in women with recurrent, ovary, fallopian tube, and primary peritoneal cancer who will be treated with a carboplatincontaining chemotherapy regimen.
  Interventions: Drug: carboplatin

INTERVENTIONS:
Drug: carboplatin — Carboplatin Standard 30-minute infusion. All patients will receive identical chemotherapy premedications including dexamethasone 20mg the night before and morning of infusion, montelukast 10mg once daily for three days prior to carboplatin infusion, and ranitidine 50mg (or famotidine 20mg IV)IV and diphenhydramine 50mg IV before carboplatin infusion.
  Arms: Standard 30-minute infusion
Drug: carboplatin — Extended 3-hour infusion carboplatin. All patients will receive identical chemotherapy premedications including dexamethasone 20mg the night before and morning of infusion, montelukast 10mg once daily for three days prior to carboplatin infusion, and ranitidine 50mg IV (or famotidine 20mg IV) and diphenhydramine 50mg IV before carboplatin infusion.
  Arms: extended 3-hour infusion

SUMMARY:
Patients who have this kind of cancer are often treated with several drugs. Carboplatin is one that seems to work for many treatment cycles. Even though it may work against the cancer, the patient can become allergic to it. If that happens, they would have to stop taking the drug. The standard way to give carboplatin is by vein over 30 minutes. Some people have been given carboplatin over 3 hours rather than 30 minutes and had fewer allergies than expected.

The purpose of this study is to:

Find out if giving carboplatin over three hours can prevent the allergy.

See if medicine given before the carboplatin can help reduce the risk of allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* MSKCC Histologically confirmed ovarian, fallopian tube or primary peritoneal carcinoma.
* Patient has received at least one prior platinum-containing (cisplatin or carboplatin) regimen
* Age ≥ 21 years old
* Karnofsky Performance Status (KPS) > or = to 70%
* Adequate hematologic, hepatic and renal function as defined below:
* Hemoglobin ≥ 7.0 g/dl
* Absolute neutrophil count ≥ 1,000/mm3
* Platelet count ≥ 100,000/mm3
* Serum creatinine ≤ 1.5 x the upper limit of normal or calculated creatinine clearance ≥ 60 mL/min

Exclusion Criteria:

* Prior carboplatin or cisplatin hypersensitivity reaction
* Uncontrolled intercurrent illness including infection, congestive heart failure, myocardial infarction, transient ischemic attack or stroke within 6 months. Any such conditions that have occurred in the last 6 months but are no longer active at the time of registration are not considered exclusionary.
* Patients receiving other investigational agents
* Patients with HIV disease will be permitted, only if they are on effective antiretroviral therapy, have a CD4 count greater than 400, and have had no opportunistic infections within the past 6 months
* Pregnant or lactating women
* Life expectancy of less than 12 weeks

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin O'Cearbhaill, MD BCh, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard 30-minute Infusion | Extended 3-hour Infusion
Started | 74 | 72
Completed | 58 | 56
Not Completed | 16 | 16
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Complete Response after 4 Cycles | 1 | 0
Not completed — Complete Response after 3 Cycles | 0 | 1
Not completed — Progression of Disease prior to 5 Cycles | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard 30-minute Infusion | Extended 3-hour Infusion | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 50 | 89
  >=65 years | 35 | 22 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 72 | 146
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 5 | 8
  White | 66 | 62 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 72 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without Hypersensitivity Reaction
Description: The primary objective of this study is to determine if patients have lower rates of hypersensitivity reactions by comparing the number of participants with and without hypersensitivity reaction
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard 30-minute Infusion | Extended 3-hour Infusion
Number analyzed (Participants) | 58 | 56
Participants
  Experienced HSR (Hypersensitivity Reaction) | 9 | 6
  Did not experience HSR (Hypersensitivity Reaction) | 49 | 50

2. Secondary Outcome: The Number of People With Successful Planned Treatment Completion of Carboplatin in Each Group
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard 30-minute Infusion | Extended 3-hour Infusion
Number analyzed (Participants) | 58 | 56
Participants
  Planned treatment completion | 49 | 50
  Planned treatment not completed | 9 | 6

3. Secondary Outcome: Perform a Cost-identification Analysis of Extended Infusion Carboplatin to Estimate the Cost Per Hypersensitivity Reaction Prevented.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Standard 30-minute Infusion | Extended 3-hour Infusion
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Odds Ratio for the Relationship of Baseline Variables to the Carboplatin Hypersensitivity Rate
Description: Perform exploratory analyses to correlate hypersensitivity rate to history of atopy, prior drug allergies, number of lifetime platinum cycles, duration since last platinum, and concomitant chemotherapy agent.
Time Frame: 2 years
Population: Among the evaluable 114 participants, 15 experienced a Hypersensitivity Reaction/HSR. 6 of the 56 participants in the extended-infusion group and 9 of the 58 participants in the standard-infusion group. These participants were analyzed as a group as the relationship of baseline variables to the rate of carboplatin HSRs were analyzed.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- Participants Who Experienced HSR: Participants who Experienced Hypersensitivity Reaction
Arm/Group | Participants Who Experienced HSR
Number analyzed (Participants) | 15
Odds Ratio
  # of Prior platinum-based regimens (>2 vs 1) | 2.5 [0.8 to 7.5]
  Prior cisplatin regimen | 1.5 [0.5 to 4.4]
  Platinum-free interval | 1 [.96 to 1]
  History of drug allergies | 0.8 [0.3 to 2.4]
  History of food allergies | 2.2 [0.5 to 9.2]
  History of atopy | 2 [0.6 to 5.8]

ADVERSE EVENTS:
Time Frame: From baseline to up to 3 months after last treatment, up to 2 years
Arm/Group | Standard 30-minute Infusion | Extended 3-hour Infusion
All-Cause Mortality (participants affected / at risk) | 57/74 | 49/72
Serious Adverse Events (participants affected / at risk) | 10/74 | 11/72
Other Adverse Events (participants affected / at risk) | 26/74 | 24/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard 30-minute Infusion (N=74) | Extended 3-hour Infusion (N=72)
Abdominal Infection (Infections and infestations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 9
Ascites (Gastrointestinal disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 6
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Infections and infestations (Infections and infestations) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard 30-minute Infusion (N=74) | Extended 3-hour Infusion (N=72)
Allergic reaction (Immune system disorders) | 9 | 7
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 7 | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 5
Resp, thoracic & mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin & subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT01248962/Prot_SAP_000.pdf